CLINICAL TRIAL: NCT05839457
Title: Safe-space Program in Secondary Schools to Address School-related Gender-based Violence in Zambia: a Cluster Randomized Controlled Trial
Brief Title: Addressing School-related Gender-based Violence as Part of the Keeping Girls in School Initiative in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Bank (Other)
Responsible Party: Principal Investigator, Wei Chang, Economist, World Bank
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: p151451
Record Dates: First submitted 2023-03-16; First posted 2023-05-03 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Gender-based Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Empowerment Pilot
  Interventions: Behavioral: Empowerment Pilot
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Empowerment Pilot — The Empowerment Pilot is a school-based program aimed to raise awareness and change attitudes around SRGBV among students and teachers and promote gender equality. This intervention includes training provided by Teacher Mentors to other teachers in school, learning sessions delivered via safe spaces for student learners, and guidance for engaging parent-teacher committees.
  Arms: Intervention group

SUMMARY:
The objective of this mixed-methods study is to evaluate the effectiveness of a school-based safe-space program delivered to secondary school students in Zambia. The quantitative component of the study uses a randomized controlled trial to measure changes in students' experience of school-related gender-based violence (SRGBV), attitudes towards gender and SRGBV, socio-emotional well-being, and school climate, among other outcomes. Meanwhile, the qualitative component of the study aims to understand the prevailing norms around SRGBV in schools, the perception of the intervention and its impact, and the potential mechanisms through which the intervention generates its outcomes.

DETAILED DESCRIPTION:
This study will evaluate the impact of the Empowerment Pilot, a school-based safe-space program delivered to secondary school students in Zambia, implemented between May and November 2023. The main question it aims to answer is whether the Empowerment Pilot changes attitudes and norms around gender roles and school-related gender-based violence (SRGBV), increases socio-emotional well-being, improves school climate, and reduces SRGBV. We use a mixed-methods triangulation design and combined qualitative and quantitative approaches in data collection and analysis to enhance the validity, depth, and relevance of our findings. Data will be collected from approximately 6,000 adolescent girls and boys and their teachers across three districts in Zambia.

The mixed-methods evaluation gives equal importance to the qualitative and quantitative components. However, this registration primarily describes the quantitative component of the study.

ELIGIBILITY:
Inclusion Criteria for Adolescent Participants:

* Students enrolled in grades 8 - 11 of secondary schools in the 2023 school year at the start of the intervention

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Experience of any SRGBV, past two weeks | two weeks prior to the endline survey
  A binary variable of self-reported experience of any SRGBV in the past two weeks
Experience of any SRGBV, past school term | ~4 months (Term 3 of School Year 2023)
  A binary variable of self-reported experience of any SRGBV in the past school term
Attitudes towards gender roles and SRGBV (adolescents) | ~4 months post-intervention
  A normalized index based on 16 items that measure attitudes towards gender roles, SRGBV, and support to victims
School climate | ~4 months post-intervention
  A composite score based on 16 statements about aspects of school climate and student-teacher interactions
Socio-emotional well-being | ~4 months post-intervention
  A normalized index based on 3 scales related to subjective well-being: perceived social support; perceived safety; and anxiety.

SECONDARY OUTCOMES:
Knowledge of SRGBV | ~4 months post-intervention
  the fraction of correct responses to 12 questions that ask whether an act is considered violence
School absenteeism | one month prior to the endline survey
  number of days an adolescent missed in the last completed month
School enrollment | ~4 months post-intervention
  A binary indicator for school enrollment status
General self-efficacy | ~4 months post-intervention
  a composite score of 10 items on the General self-efficacy scale.
Assertive communication | ~4 months post-intervention
  a composite score of 6 items on the Assertiveness Communication scale
Gender equitable injunctive norms | ~4 months post-intervention
  A composite score of injunctive norms for gender equality norms, GBV, Corporal punishment, and GBV reporting
Gender equitable descriptive norms | ~4 months post-intervention
  A composite score of descriptive norms for gender equality, GBV, Corporal punishment, and GBV reporting
Experience of sexual violence, past two weeks | 2 weeks prior to the endline survey
  A binary variable of self-reported experience of any type of sexual violence reported by the respondent
Experience of emotional violence, past two weeks | 2 weeks prior to the endline survey
  A binary variable of self-reported experience of any type of emotional violence reported by the respondent
Experience of physical violence, past two weeks | 2 weeks prior to the endline survey
  A binary variable of self-reported experience of any type of physical violence reported by the respondent
Experience of sexual violence, past school term | ~4 months (Term 3 of School Year 2023)
  A binary variable of self-reported experience of any type of sexual violence reported by the respondent
Experience of emotional violence, past school term | ~4 months (Term 3 of School Year 2023)
  A binary variable of self-reported experience of any type of emotional violence reported by the respondent
Experience of physical violence, past school term | ~4 months (Term 3 of School Year 2023)
  A binary variable of self-reported experience of any type of physical violence reported by the respondent
Attitudes towards gender roles and norms | ~4 months post-intervention
  a composite score based on 7 items with a likert-scale
Attitudes towards SRGBV | ~4 months post-intervention
  a composite score based on 7 items with a likert-scale
Attitudes towards reporting SRGBV | ~4 months post-intervention
  a composite score based on 2 items with a likert-scale
Bystander reporting | ~4 months post-intervention
  A binary indicator coded to 1 if adolescent reported any case of violence in the past school term (0/1)
Attitudes towards bystander intervention (vignettes) | ~4 months post-intervention
  A score based on 2 questions on attitudes towards bystander intervention in hypothetical situations
Descriptive norms around bystander intervention (vignettes) | ~4 months post-intervention
  A score based on 2 questions on descriptive norms
Injunctive norms around bystander intervention (vignettes) | ~4 months post-intervention
  A score based on 2 questions on injunctive norms
Aspiration - education attainment | ~4 months post-intervention
  a variable that indicates the level of formal education the respondent would like to complete
Aspiration for a career | ~4 months post-intervention
  a binary indicator coded to 1 if adolescent aspires for professional career
Perceived social support | ~4 months post-intervention
  mean score based on the Multidimensional Scale of Perceived Social Support
Anxiety | ~4 months post-intervention
  a composite score based on GAD-7 anxiety scale (Spitzer et al., 1999)
Perceived safety at school | ~4 months post-intervention
  A composite score of 5 items about whether respondent feels safe at school
Aspired age of marriage | ~4 months post-intervention
  a binary indicator coded to 1 if adolescent aspires to marry after the age of 18
Agency | ~4 months post-intervention
  A composite score based on 20 items that measure different aspects of agency, including freedom of movement, voice, behavioral control and decision making, adapted from the Agency Scale from the Global Early Adolescent Study (Zimmerman et al., 2019)

OTHER OUTCOMES:
Teachers' knowledge of SRGBV | ~4 months post-intervention
  the fraction of correct responses to 12 questions that ask whether an act is considered violence
Teachers' assessment of school climate | ~4 months post-intervention
  An index based on 17 items that measure to what extent the school climate is safe for both boys and girls
Attitudes towards gender roles and SRGBV (teachers) | ~4 months post-intervention
  A normalized index based on 16 items that measure attitudes towards gender roles, SRGBV, and support to victims

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chang, Principal Investigator — World Bank
Locations (1):
- secondary schools in Kasama, Mpongwe, and Zambezi districts, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No